CLINICAL TRIAL: NCT02273570
Title: Single-center, Open-label, Randomized Study of Anemia Management Improvement in End Stage Renal Disease (ESRD) Patients With Secondary Hyperparathyroidism
Brief Title: Optimal Anemia Treatment in End Stage Renal Disease (ERSD)
Acronym: OPTIMAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Sant'Anna (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AOSantAnna
Record Dates: First submitted 2014-06-27; First posted 2014-10-24 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: Hyperparathyroidism, Secondary; Anemia; Vascular Stiffness; Vascular Calcification
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Anemia; Vascular Calcification | interventions — Standard of Care; calcium acetate; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): Control group: standard care. The iPTH target in this group is 300-540 pg/ml
  Interventions: Drug: standard care
- Optimal CKD-MBD control (Experimental): Optimal CKD-MBD control: in this group the PTH target is150-300 pg/ml to be achieved with a therapeutic algorithm
  Interventions: Drug: Optimal (I. iPTH control: Zemplar®,Mimpara®; phosphorous control: Renvela®, Phoslo®, Osvaren®, Foznol®,Maalox®; calcium control: calcium and vitamin D

INTERVENTIONS:
Drug: standard care — Standard care. Patients allocated to this study arm will be treated with all drugs available for PTH control (at the investigator discretion) to obtain a iPTH of 300-540 pg/ml.
  Other Names: Drugs available on the market control iPTH
  Arms: control
Drug: Optimal (I. iPTH control: Zemplar®,Mimpara®; phosphorous control: Renvela®, Phoslo®, Osvaren®, Foznol®,Maalox®; calcium control: calcium and vitamin D — Optimal care. Patients allocated to this study arm will be treated with all drugs available for PTH control (at the investigator discretion - see therapeutic algorithm) to obtain a iPTH of less than 300 pg/ml.
  Other Names: Drugs available on the market control iPTH
  Arms: Optimal CKD-MBD control

SUMMARY:
Clinical study aimed at improving anemia management in End Stage Renal Disease Patient (ESRD) on maintenance Hemodialysis with evidence of Chronic Kidney disease Mineral Bone Disorder (CKD-MBD)

DETAILED DESCRIPTION:
Anemia is one of the most worrisome complications of Chronic Kidney Disease (CKD). Numerous prospective studies have repeatedly documented an increase risk of morbidity and mortality associated with lower levels of hemoglobin (Hb). Hence the international guidelines on patient care suggest the use of Erythropoietin Stimulating Agents (ESA), iron, folates supplementation for anemia correction.

However, recent randomized controlled trials (RCT) have demonstrated that hemoglobin correction to normal levels increases the risk of major cardiovascular (CV) events. Though, the reasons are still unclear, the cumulative ESA dose may at least partly explain these findings suggesting limiting ESA to the minimal dose allowed to achieve the suggested Hb targets in ESRD patients.

Among other factors, CKD-MBD has been repeatedly associated with poor more severe anemia and higher dose of ESA. However, the latest Kidney Disease: Improving Global Outcomes (KDIGO) guidelines on CKD-MBD management suggest a higher reference target for intact parathyroid hormone (iPTH) (2-9 fold the upper level of the normal range) when compared to the National Kidney Foundation (NKF) guidelines published in 2003 (150-300 pg/ml).

A few observational studies suggest a linear inverse association between intact iPTH and ESA dose even for iPTH value within the iPTH target level proposed by the KDIGO working group. Similarly, a large body of evidence supports the notion that the higher the iPTH the faster the CV system deterioration in ESRD.

Aim of the study is to test whether a tighter iPTH control to achieve a iPTH level lower than 300 pg/ml vs iPTH levels between 300-540 pg/ml is associated with a ESA dose reduction and a slower CV system deterioration in ESRD patients receiving dialysis.

STUDY DESIGN Pilot, single center, open label with blinded end point (PROBE-Prospective Randomized Open Blinded End-Point) aimed at improving patient care.

Eligible patients will be randomized (1:1) to either:

(A) Control group: standard care. The iPTH target in this group is 300-540 pg/ml (B) Optimal CKD-MBD control: in this group the iPTH target is150-300 pg/ml to be achieved with a therapeutic algorithm.

TREATMENTS

All patients will be randomized (1:1) to either:

(A) Control group: standard care. The iPTH target in this group is 300-540 pg/ml.

(B) Optimal CKD-MBD control:: in this group the iPTH target is 150-300 pg/ml to be achieved with a therapeutic algorithm:

I. iPTH control: in order to achieve the iPTH target (150-300 pg/ml), all patients will receive 400 IU/day of vitamin-25-OH-D (25OHD) and a flexible dose of any active vitamin D available in Italy (calcitriol and paricalcitol-"Zemplar®") at the maximum dose of 6 mcg/week of paricalcitol("Zemplar®")of equivalent (see existing conversion table). Patients will also receive a flexible dose of cinacalcet("Mimpara®") to a maximum dose of 90 mg/day.

II. Phosphorous control: all patients need to achieve a serum phosphorous level lower than 5.5 mg/dl. All available phosphate binders are allowed [sevelamer("Renvela®"), calcium carbonate, calcium acetate("Phoslo®"), calcium acetate/magnesium carbonate ("Osvaren®"), lanthanum carbonate "Foznol®"). A rescue therapy with aluminum("Maalox®") is allowed for no more than 30 days.

III. Serum calcium control: the suggested target is less than 9.5 mg/dl. In case of serum calcium greater than 9.5 mg/dl the calcium and vitamin D dose should be lowered in order to lower the risk of vascular calcification deposition and progression

ELIGIBILITY:
INCLUSION CRITERIA.

* Men and women
* Age >18 years
* Maintenance dialysis via Artero-Venous fistula
* ESA use
* iPTH between 300-600 pg/ml
* Hb between 10.0-11.5
* Kt/V greater/equal than 1.2
* Signed informed consent prior to the initiation of the study

EXCLUSION CRITERIA: None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
percent reduction in weekly ESA consumption to maintain Hb levels within the recommended range 10.0-11.5 g/dl | baseline and after 12 months of followup
  Primary objective: to test whether a tighter PTH control to achieve a PTH level lower than 300 pg/ml vs PTH levels between 300-540 pg/ml is associated with a lower ESA dose use to achieve the target Hb of 10.0-11.5 g/dl

SECONDARY OUTCOMES:
Change in iron status and storage. | baseline and after 12 months of followup
  Secondary objective: to test whether a tighter PTH control to achieve a PTH level lower than 300 pg/ml vs PTH levels between 300-540 pg/ml is associated with a better iron storage and mobilization.
Difference in prevalence of cardiac valvular calcification progression detected by echocardiography between groups. | baseline and after 12 months of followup
  Secondary objective: to test whether a tighter PTH control to achieve a PTH level lower than 300 pg/ml vs PTH levels between 300-540 pg/ml is associated with cardiac valves deposition and progression attenuation.
Difference in pulse wave velocity assessed by applanation tonometry between groups. | baseline and after 12 months of followup
  Secondary objective: to test whether a tighter PTH control to achieve a PTH level lower than 300 pg/ml vs PTH levels between 300-540 pg/ml is associated with arterial stiffness increase attenuation
CKD-MBD control | baseline and after 12 months of followup
  Secondary objective: to test whether a tighter PTH control to achieve a PTH level lower than 300 pg/ml vs PTH levels between 300-540 pg/ml is associated with a better CKD-MBD control

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Bellasi, MD, Principal Investigator — Azienda Ospedaliera Sant'Anna, Ospedale Sant'Anna-Como
Locations (1):
- Azienda Ospedaliera Sant'Anna, San Fermo Della Battaglia (CO), Italy

REFERENCES:
- [Background] Capuano A, Serio V, Pota A, Memoli B, Andreucci VE. Beneficial effects of better control of secondary hyperparathyroidism with paricalcitol in chronic dialysis patients. J Nephrol. 2009 Jan-Feb;22(1):59-68. PMID 19229819
- [Background] Ebben JP, Gilbertson DT, Foley RN, Collins AJ. Hemoglobin level variability: associations with comorbidity, intercurrent events, and hospitalizations. Clin J Am Soc Nephrol. 2006 Nov;1(6):1205-10. doi: 10.2215/CJN.01110306. Epub 2006 Sep 6. PMID 17699349
- [Background] Fishbane S, Berns JS. Hemoglobin cycling in hemodialysis patients treated with recombinant human erythropoietin. Kidney Int. 2005 Sep;68(3):1337-43. doi: 10.1111/j.1523-1755.2005.00532.x. PMID 16105069
- [Background] Gilbertson DT, Ebben JP, Foley RN, Weinhandl ED, Bradbury BD, Collins AJ. Hemoglobin level variability: associations with mortality. Clin J Am Soc Nephrol. 2008 Jan;3(1):133-8. doi: 10.2215/CJN.01610407. Epub 2007 Nov 28. PMID 18045862
- [Background] Lacson E Jr, Ofsthun N, Lazarus JM. Effect of variability in anemia management on hemoglobin outcomes in ESRD. Am J Kidney Dis. 2003 Jan;41(1):111-24. doi: 10.1053/ajkd.2003.50030. PMID 12500228
- [Background] Pisoni RL, Bragg-Gresham JL, Young EW, Akizawa T, Asano Y, Locatelli F, Bommer J, Cruz JM, Kerr PG, Mendelssohn DC, Held PJ, Port FK. Anemia management and outcomes from 12 countries in the Dialysis Outcomes and Practice Patterns Study (DOPPS). Am J Kidney Dis. 2004 Jul;44(1):94-111. doi: 10.1053/j.ajkd.2004.03.023. PMID 15211443
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Work Group. KDIGO clinical practice guideline for the diagnosis, evaluation, prevention, and treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl. 2009 Aug;(113):S1-130. doi: 10.1038/ki.2009.188. PMID 19644521
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for bone metabolism and disease in chronic kidney disease. Am J Kidney Dis. 2003 Oct;42(4 Suppl 3):S1-201. No abstract available. PMID 14520607